CLINICAL TRIAL: NCT00355498
Title: Amyloid Plaque and Tangle Imaging in Aging and Dementia
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gary Small, MD, Professor, University of California, Los Angeles
Other Study IDs: IA0093; P01AG025831-01 (NIH); P01-AG024831-01
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Memory Disorders; Alzheimer's Disease
Keywords: functional magnetic resonance imaging; positron emission tomography; beta-amyloid; tau
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Plaque, Amyloid; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Controls
- 2: Mild Cognitive Impairment
- 3: Alzheimer's disease
- 4: FTD

SUMMARY:
Amyloid senile plaques (SPs) and neurofibrillary tangles (NFTs) are neuropathological hallmarks of Alzheimer's disease (AD) that also accumulate in key brain regions in association with normal aging. This project will expand an established program in early detection and prevention of AD designed (1) to identify presymptomatic persons most likely to benefit from early intervention and (2) to provide an objective, noninvasive means to monitor therapeutic trials.

DETAILED DESCRIPTION:
A total of 165 volunteers will be recruited for this 2-year study. Participants will receive a baseline clinical and imaging evaluation and one follow-up evaluation two years later. These evaluations will include clinical and neuropsychological assessments, structural MRI and/or PET scans. Additional scans and scanning procedures will be performed on a subset of participants and participant visits, including serotonin density levels.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in a clinical and brain imaging study
* Age 30 years or older
* No significant cerebrovascular disease - modified Ischemic Score of ≤ 4
* For volunteers with MCI or dementia, there must be a family member or potential caregiver available
* Adequate visual and auditory acuity to allow neuropsychological testing
* Screening laboratory tests and ECG without significant abnormalities that might interfere with the study.

Exclusion Criteria:

* Evidence of neurologic or other physical illness that could produce cognitive deterioration; in addition to a physical and neurological examination, volunteers will be screened for Parkinson's disease
* History of myocardial infarction within the previous year or unstable cardiac disease
* Uncontrolled hypertension (systolic BP>170 or diastolic BP>100), history of significant liver disease, clinically significant pulmonary disease, diabetes, or cancer
* Major psychiatric disorders, such as bipolar disorder or schizophrenia
* Because medications can affect cognitive functioning, volunteers needing medicines that could influence psychometric test results will be excluded; use of any of the following drugs will also exclude volunteers: centrally active beta-blockers, narcotics, clonidine, anti-Parkinsonian medications, benzodiazepines, systemic corticosteroids, and medications with significant cholinergic or anticholinergic effects, anti-convulsants, or warfarin
* Current diagnosis or history of alcoholism or drug dependence
* Evidence of untreated depression as determined by a HAM-D (Hamilton, 1960) score of ≥ 12 (17-item version) or untreated anxiety by a score of ≥ 8 on the Hamilton Anxiety Scale (HAM-A; Hamilton, 1959)
* Use of any investigational drugs within the previous month or longer, depending on drug half-life
* Contraindication for MRI scan (e.g., metal in body, claustrophobia)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is selected from UCLA primary care clinics, UCLA memory clinic, residents from the California counties of Orange and Los Angeles who answer ads placed in newspapers in these areas.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2005-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary W. Small, MD, Principal Investigator — University of California, Los Angeles, Neuropsychiatric Institute
Locations (1):
- Jane & Terry Semel Institute for Neuroscience & Human Behavior, Los Angeles, California, United States

REFERENCES:
- [Background] Ercoli L, Siddarth P, Huang SC, Miller K, Bookheimer SY, Wright BC, Phelps ME, Small G. Perceived loss of memory ability and cerebral metabolic decline in persons with the apolipoprotein E-IV genetic risk for Alzheimer disease. Arch Gen Psychiatry. 2006 Apr;63(4):442-8. doi: 10.1001/archpsyc.63.4.442. PMID 16585474
- [Background] Kepe V, Barrio JR, Huang SC, Ercoli L, Siddarth P, Shoghi-Jadid K, Cole GM, Satyamurthy N, Cummings JL, Small GW, Phelps ME. Serotonin 1A receptors in the living brain of Alzheimer's disease patients. Proc Natl Acad Sci U S A. 2006 Jan 17;103(3):702-7. doi: 10.1073/pnas.0510237103. Epub 2006 Jan 9. PMID 16407119
- [Background] Small GW, Silverman DH, Siddarth P, Ercoli LM, Miller KJ, Lavretsky H, Wright BC, Bookheimer SY, Barrio JR, Phelps ME. Effects of a 14-day healthy longevity lifestyle program on cognition and brain function. Am J Geriatr Psychiatry. 2006 Jun;14(6):538-45. doi: 10.1097/01.JGP.0000219279.72210.ca. PMID 16731723
- [Derived] Merrill DA, Siddarth P, Raji CA, Emerson ND, Rueda F, Ercoli LM, Miller KJ, Lavretsky H, Harris LM, Burggren AC, Bookheimer SY, Barrio JR, Small GW. Modifiable Risk Factors and Brain Positron Emission Tomography Measures of Amyloid and Tau in Nondemented Adults with Memory Complaints. Am J Geriatr Psychiatry. 2016 Sep;24(9):729-37. doi: 10.1016/j.jagp.2016.05.007. Epub 2016 May 13. PMID 27421618